CLINICAL TRIAL: NCT06853834
Title: Prospective Randomized Controlled Study Comparing Diagnostic Yield of Endobronchial Cryo Biopsy vs Forceps Biopsy in Patients Undergoing Endobronchial Ultrasound Guided Transbronchial Needle Aspiration for Suspected Sarcoidosis
Brief Title: Comparative Diagnostic Yield of Endobronchial Cryo Biopsy vs Forceps Biopsy in Patients With Suspected Sarcoidosis
Acronym: CREBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Ajmal Khan, Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DMEBBRCT001
Record Dates: First submitted 2025-02-24; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Sarcoidosis Lung; Pulmonary Sarcoidosis
Keywords: Forceps Endobronchial Biopsy; Cryo-Endobronchial Biopsy; Pulmonary Sarcoidosis; Diagnostic yield of endobronchial biopsy in sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant
Masking Description: Pathologist examining the sample will be blinded for the type of forceps vs cryo biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryo-Endobronchial Biopsy (Experimental): Endobronchial biopsy obtained using CRYO-Probe
  Interventions: Device: Cryobiopsy with liquid nitrogen
- Forceps Endobronchial Biopsy (Active Comparator): Endobronchial Biopsy using Standard Bronchoscopic Biopsy Forceps
  Interventions: Device: Endobronchial Forceps Biopsy

INTERVENTIONS:
Device: Cryobiopsy with liquid nitrogen — Forceps vs Cryo Endobronchial Biopsy
  Other Names: Forceps biopsy; Cryo Biopsy
  Arms: Cryo-Endobronchial Biopsy
Device: Endobronchial Forceps Biopsy — Comparision of forceps and cryo endobronchial biopsy
  Other Names: Cryo Biopsy; Forcpes Biopsy
  Arms: Forceps Endobronchial Biopsy

SUMMARY:
Sarcoidosis is a multi-systemic granulomatous disease of unknown cause that is characterized by the formation of non-caseous epithelioid cell granulomas. Sarcoidosis involves the respiratory system in > 90% of cases, usually the hilar and mediastinal nodes, and, less frequently, the lung tissue. Airway involvement, as judged by clinical features, physiologic testing, imaging techniques, bronchoscopy, and airway mucosal biopsy, has been observed in nearly two-thirds of patients with sarcoidosis. Although sarcoidosis involving thoracic lymph nodes and pulmonary parenchyma is familiar to most clinicians, airway involvement is often overlooked. The frequency of airway involvement increases as the parenchymal disease progresses, and\airway involvement is associated with increased morbidity, respiratory symptoms, and mortality. The initial airway abnormality is the inflammation manifested by mucosal edema, erythema, and the formation of granulomas. As the airway disease progresses, the mucosa may demonstrate granularity, nodularity, cobble stoning, and friability. Sarcoid granulomas tend to develop along the bronchovascular bundle or in the vicinity of the airways. Overall quality of the endobronchial biopsy (EBB) will depend on the method by which it is obtained and cryo-EBB will most likely to provide better tissue for the diagnosis in comparison to forceps biopsy which has smaller sample as well as crush artifacts. Therefore, it is hypothesized that cryo-EBB will be better than forceps EBB and combined together it will increase the overall diagnostic yield of the sarcoidosis when combined with lymph node sampling by endobronchial ultrasound guided trans-bronchial needle aspiration (EBUS-TBNA).

1. Primary objective: To compare the diagnostic yield of cryo-EBB with forceps biopsy in patients undergoing routine EBUS-TBNA for suspected sarcoidosis.
2. Secondary Objective: To evaluate the overall diagnostic yield of combined endobronchial biopsy and EBUS-TBNA in patients undergoing routine EBUS-TBNA for suspected sarcoidosis.

The relevance and the expected outcome of the proposed study

1. The study will provide insight to obtain an endobronchial biopsy either with cryo probe or forceps
2. The study will also provide information regarding overall increase in diagnostic yield if any when the endobronchial biopsies are combined with EBUS-TBNA.

DETAILED DESCRIPTION:
The study will consist of consecutive patients undergoing routine EBUS-TBNA for suspected sarcoidosis AND subsequently confirmed on clinical, radiology and non-caseating granuloma on histopathology. .

150 patients will be randomized into either cryo-EBB or forceps biopsy from a computer-generated randomized table. 75 patients will be included in each arm.

Determination of the sample size was based on the primary outcome of the proportion of diagnostic yield between two independent groups. Using the z test of proportion for two independent samples to detect a one-sided target difference between the groups of 15% with 85% power and a level of significance of 5%, each group required 69 participants. With an expected attrition rate of 8-10%, we capped the total number of participants in each arm of the study at 75.

Subsequent to EBUS-TBNA, video bronchoscopy will be performed to obtain the endobronchial biopsy by using either forceps or cryo-proble. Three endobronchial biopsies from primary carina and both left and right secondary carina will be taken in each patients irrespective of the endobronchial abnormality. Additional biopsies will be taken from any endobronchial abnormality detected during the examination.

The biopsy samples will be fixed in neutral 10% buffered formalin. In the pathology laboratory the sample will be embedded in paraffin followed by staining with hematoxylin and eosin or special stain according to the requirement to allow an exact classification. The samples will be analyzed and assessed by one pathologist according to common standards describing adequacy of the sample, crush artifacts, specific diagnosis. The pathologist will be blinded from the biopsy technique that has been used.

Diagnostic yield will be defined by the ability to make an adequate diagnosis on histopathological examination of the sampled tissue. Diagnostic yield will be calculated for each biopsy technique as the number of diagnostic procedures divided by number of non-diagnostic procedures plus the number of diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

All patients of suspected pulmonary sarcoidosis scheduled for routine EBUS-TBNA

Exclusion Criteria:

1. Patient age less than 18 years
2. Patients with co-morbid conditions like Diabetes mellitus, renal failure, chronic liver disease or any other chronic disease.
3. Patients already on treatment with steroids or h/o steroids intake in last three months or on disease modifying and immunosuppressive drugs.
4. Final Diagnosis other than sarcoidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield | Two week after the end of enrollment
  To compare the diagnostic yield of cryo-endobronchial biopsy with forceps biopsy in patients undergoing routine EBUS-TBNA for suspected sarcoidosis.

SECONDARY OUTCOMES:
Over all diagnostic yield | Two week after the end of enrollment
  Overall diagnostic yield - TBNA + Endobronchial Biopsy
Complications | From enrollment to Two week after the end of enrollment
  Complications of endobronchial biopsy
Dignostic yield based on endobronchial abnormality | Two week after the end of enrollment
  Diagnostic yield in normal vs abnormal endobronchial fingins

CONTACTS AND LOCATIONS:
Overall Officials: Ajmal Khan, MBBS, MD, DM, Principal Investigator — SGPGIMS
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided
Available on request to principle investigator